CLINICAL TRIAL: NCT02306668
Title: Microbiome Analysis of the Ocular Surface in Dry Eye Disease
Brief Title: Ocular Surface Dry Eye Microbiome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Russell Van Gelder, Professor and Chair, Department of Ophthalmology, University of Washington
Other Study IDs: 46093-B
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Dry Eyes
Keywords: Dry eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Conjunctival swabs
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ocular surface discomfort: There are no interventions with this observational study

SUMMARY:
The investigators seek to characterize the identity of all microorganisms residing on the eye's surface (conjunctiva) in healthy eyes and those with dry eye syndrome, using a combination of analyses. Dry eye disease is thought to have an inflammatory basis and in the vast majority of cases the cause of the chronic inflammatory condition is unknown.

ELIGIBILITY:
Inclusion Criteria:

* dry eye syndrome with OSDI score greater than 60
* control group with OSDI score less than 30

Exclusion Criteria:

* recent history of contact lens wear
* use of topical antibiotics or prescription eye medication in past 6 months
* penetrating ocular surgery in the last 12 months
* age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit 40 subjects from University of Washington Medicine Eye Institute with ocular surface discomfort consistent with dry eye syndrome, and 40 control subjects
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Identification of bacteria or fungus from conjunctival swab | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Russell Van Gelder, MD, PhD, Principal Investigator — UW Medicine Eye Institute
Locations (1):
- UW Medicine Eye Institute, Seattle, Washington, United States